CLINICAL TRIAL: NCT02612844
Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneous NNC0143-0406 A 0.6 mmol/L in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1406-4209; 2014-005334-63 (EudraCT Number); U1111-1164-6630 (Other: WHO)
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC0143-0406 (Experimental)
  Interventions: Drug: NNC0143-0406; Drug: insulin aspart
- Insulin Aspart (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: NNC0143-0406 — Subject will receive one single dose only Subcutanesously (s.c., under the skin)
  Arms: NNC0143-0406
Drug: insulin aspart — Subject will receive one single dose only. Subcutanesously (s.c., under the skin)

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the Safety, Tolerability,Pharmacokinetics (the exposure of the trial drug in the body) and Pharmacodynamics (the effect of the investigated drug on the body) of subcutaneous NNC0143-0406 A 0.6 mmol/L in Subjects with Type 1 Diabetes

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18-55 years (both inclusive) at the time of signing informed consent
* Subjects diagnosed (clinically) with type 1 diabetes mellitus at least 365 days prior to the day of screening
* Body mass index between 18.5 and 28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products.
* Males who are sexually active and not surgically sterilised (vasectomy or otherwise) and their partners that are not using a highly effective contraception method, from randomisation until 90 days after dosing, such as double barrier contraception (e.g. condom and spermicide) or combination of either an oral contraceptive, a contraceptive patch, a diaphragm or intrauterine device, together with a physical barrier such as condom. Malesubjects must also agree to refrain from sperm donation from randomisation until 90 days after dosing
* History or presence of any clinically relevant respiratory, metabolic (including dyslipidaemia), renal, hepatic, gastrointestinal, endocrinological conditions (except conditions associated with diabetes mellitus)
* Subject who has donated any blood or plasma in the past month or more than 500 mL within 90 days prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day) who is not able or willing to refrain from smoking or use of nicotine gum or transdermal nicotine patches during the in-patient period
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event during the past 180 days) or hypoglycaemic unawareness as judged by the investigator or hospitalisation for diabetic ketoacidosis within the last 180 days

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The number of treatment emergent adverse events | From the time of dosing (Visit 2,Day 1) and until completion of the post-treatment follow-up visit (Visit 3) i.e. 11-13 days.

SECONDARY OUTCOMES:
Area under the serum NNC0143-0406 concentration-time curve | From 0 to 24 hours
Area under the glucose infusion rate-time curve | From 0 to 24 hours
The maximum glucose infusion rate | From 0 to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com